CLINICAL TRIAL: NCT02698813
Title: Safety Study of Filler Agent Composed of Umbilical Cord Mesenchymal Stem Cells and Hyaluronic Acid
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South China Research Center for Stem Cell and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCMSC-HA-1
Record Dates: First submitted 2016-02-04; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Senescence Wrinkles, Acne, Pitting Scar
MeSH Terms: conditions — Acne Vulgaris | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UCMSCs-HA (Experimental): Multipoint of Transdermal injection into the wrinkles. Injectable filler agent composed of umbilical cord mesenchymal stem cells (UCMSCs) and hyaluronic acid (HA).
  Interventions: Biological: umbilical cord mesenchymal stem cells and hyaluronic acid
- Control (Active Comparator): Procedure: Transdermal injection of hyaluronic acid only.
  Interventions: Drug: hyaluronic acid

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells and hyaluronic acid
  Arms: UCMSCs-HA
Drug: hyaluronic acid
  Arms: Control

SUMMARY:
The overall goal of this study is to evaluate the safety and exploratory efficacy of the injectable filler agent composed of umbilical cord mesenchymal stem cells and hyaluronic acid for the improvement of wrinkles, acne, pitting scar and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years;
2. Have ability to understand and comply with the study requirements, and provide the written informed consent prior to any procedures ;
3. Suitable for the medical history and physical examination like the following preoperative laboratory tests results: complete blood count, coagulation, biochemistry, electrocardiogram, hepatogram and β-human chorionic gonadotropin (hCG) for women of childbearing age.

Exclusion Criteria:

1. Patients unable to undergo surgery liposuction with Klein technique as those with severe cardiovascular disease, severe coagulation disorders including thrombophilia and pregnancy;
2. Have history or active dermal diseases, inflammation, or any related disease;
3. Had invasive aesthetic treatments or surgeries history 6 months before the treatments;
4. Had physical or chemical aesthetic treatments 1 months before the study starts;
5. Have a known history of allergic reactions like hypersensitivity to hyaluronic acid;
6. Patients with limited understanding of the procedure or have poor compliance with the study or follow-up schedule;
7. Pregnant or lactating;
8. Use of drugs;
9. Patients with preoperative results considered inadequate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with non-serious and serious adverse events | Change from baseline up to week 12 after injection.

SECONDARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) Evaluation | Change from baseline at week 2, 6 and 12.
  An improvement was judged by the outcome of the preoperative grade minus the postoperative grade in accordance with the Wrinkle Severity Rating Scale (WSRS).The severity was measured using the Wrinkle Severity Rating Scale (WSRS), where 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Extreme, which is an ordinal scale.
Global Aesthetic Improvement Scale (GAIS) Evaluation | Change from baseline at week 2, 6 and 12.
  An improvement was judged by the outcome of the preoperative grade minus the postoperative grade in accordance with the Global Aesthetic Improvement Scale (GAIS).